CLINICAL TRIAL: NCT04397978
Title: Local Ablative Therapy for Patients With Multiple (4-10) Brain Metastases
Acronym: LAT-MUM
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S63789
Record Dates: First submitted 2020-05-11; First posted 2020-05-21 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Brain Metastases, Adult
Keywords: Stereotactic radiotherapy; Brain metastases; Multiple (4-10)
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Stereotactic radiotherapy — Local ablative therapy with SRT
  Other Names: SRT

SUMMARY:
To observe the quality of life (QOL) and to report on toxicity and outcome parameters after the (repeated) use of local ablative therapy (LAT) i.e. stereotactic radiotherapy (SRT) for patients with multiple (4-10) brain metastases

DETAILED DESCRIPTION:
Phase IV prospective non-randomized observational trial (registry trial) for patients with a DS-GPA > 1.5 or an estimated life expectancy of >3 months and an established diagnosis on dedicated brain MRI of 4-10 BM of any solid primary tumor.

We plan to deliver a local ablative therapy (LAT) i.e. SRT in 1 to 5 fractions on visible BM and post-surgical cavities if applicable.

Our primary aim is to provide quality of life (QOL) data and our secondary aim is to report on several toxicity and outcome parameters for this patient cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age
2. Minimal 4 and up to a maximum of 10 synchronous BM diagnosed on a high resolution contrast-enhanced MRI scan (T1 gadolinium) not dated more than 4 weeks prior to inclusion.
3. Maximal lesion diameter of single gross tumor volume (GTV) of 3 cm
4. Maximal cumulative GTV (+CTV for cavity) of 30cm3
5. Karnofsky performance status ≥ 70
6. DS-GPA or expected overall survival (if no DS-GPA applicable) of ≥ 1.5 or >3 months respectively.
7. Any solid primary tumour. Lymphoma, germ cell tumor, small cell lung carcinoma and multiple myeloma are excluded.
8. Ability to provide written informed consent and to participate in the procedure of the questionnaires.

Exclusion Criteria:

1. BM not amenable to SRT
2. Previous SRT or surgery on the same lesion
3. Co-morbidities considered clinically precluding the safe use of an MRI examination or SRT
4. Any psychological, sociological or geographical issue potentially hampering compliance with the study
5. Pregnancy
6. Concurrent use of systemic therapy
7. More than 10 BM on planning-MRI
8. Maximum cumulative GTV (+CTV for cavity) of more than 30cm3 on planning-MRI
9. A brainstem metastasis with a PTV of more than 20 cm3
10. Leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with an established diagnosis on dedicated brain magnetic resonance (MRI) of 4-10 brain metastases (BM) of any solid tumor with an estimated life expectancy of >3 months or a disease specific grade prognostic index (DS-GPA) of ≥ 1.5.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life | From baseline to 3 month after radiotherapy
  Measured by the EQ-5D-5L questionnaire
Quality of life | From baseline to 3 month after radiotherapy
  Measured by the QLQ-BN20 questionnaire
Quality of life | From baseline to 3 month after radiotherapy
  Measured by the PRO-CTCAE

SECONDARY OUTCOMES:
Quality of life | From baseline to 1,6,9 and 12 month (+q3month) after radiotherapy
  Measured by the EQ-5D-5L questionnaire
Quality of life | From baseline to 1,6,9 and 12 month (+q3month) after radiotherapy
  Measured by the QLQ-BN20 questionnaire
Quality of life | From baseline to 1,6,9 and 12 month (+q3month) after radiotherapy
  Measured by the PRO-CTCAE
Local control | Time from SRT until local progression or death whichever comes first, up to 3 years after LAT
  Local control of the irradiated metastases
Survival | Time from SRT until the occurrence of new brain metastases or death whichever comes first, up to 3 years after LAT
  Brain metastasis free survival
Survival | Time from SRT until death from any cause
  Overall survival
Radiotherapy induced toxicity | From baseline to ≤ 90 days after radiotherapy
  Acute toxicity
Radiotherapy induced toxicity | From > 90 days after radiotherapy through study completion
  Late toxicity
Radiotherapy induced toxicity | Change in toxicity measured from baseline up to 3 years after radiotherapy
  Occurrence of radionecrosis

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Berkovic, MD, Principal Investigator — UZ Leuven; Maarten Lambrecht, PHD, Study Chair — UZ Leuven; Eva Oldenburger, MD, Study Chair — UZ Leuven; An Nulens, Study Chair — UZ Leuven; Lien Smets, BA, Study Chair — UZ Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No